CLINICAL TRIAL: NCT07269977
Title: mSCI: mHealth for Supporting Psychosocial Health of Military Service Members With SCI and Their Family Caregivers
Brief Title: mSCI: Mobile Health App for Veterans With SCI and Caregivers
Status: Recruiting | Type: Observational
Sponsor: University of Pittsburgh (Other)
Collaborators: Congressionally Directed Medical Research Programs (U.S. Federal Agency)
Responsible Party: Principal Investigator, Yong Choi, Assistant Professor, University of Pittsburgh
Other Study IDs: STUDY24030058; HT94252410748 (Other Grant/Funding Number: US Army Medical Research and Materiel Command (USAMRMC)); CDMRP-SC230134 (Other Grant/Funding Number: Congressionally Directed Medical Research Programs)
Record Dates: First submitted 2025-11-20; First posted 2025-12-08 (Actual); Last update posted 2025-12-12 (Actual); Status verified 2025-12

CONDITIONS: Spinal Cord Injuries (SCI); Spinal Cord Injury; Spinal Cord Injuries (Complete and Incomplete); Family Caregivers; Families of Veterans; Disabled Veterans
Keywords: Spinal Cord Injury; Veterans; Veterans with SCI; SCI; SCI/D; Spinal Cord Injuries; Spinal Cord Disorder; Family caregiver; Primary caregiver; mobile health app; smartphone app; Imhere; Veterans support; paralyzed veterans; disabled veterans; mobile health support; mobile health; telemedicine
MeSH Terms: conditions — Spinal Cord Injuries; Spinal Cord Diseases

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Veterans with SCI: Veterans with Spinal Cord Injury
  Interventions: Other: iMHERE 2.0. A mobile health App designed to support veterans with SCI manage their self care, and their caregivers
- Primary Caregivers of Veterans with SCI: Family member who is the main (primary) caregiver of the veterans with SCI
  Interventions: Other: iMHERE 2.0. A mobile health App designed to support veterans with SCI manage their self care, and their caregivers

INTERVENTIONS:
Other: iMHERE 2.0. A mobile health App designed to support veterans with SCI manage their self care, and their caregivers — iMHere is a mobile health technology designed to support veterans with SCI and their caregivers.

SUMMARY:
Caregivers of persons with Spinal Cord Injury (SCI) face increased risk of psychological distress, health problems, reduced quality of life, relationship strain, and restrictions in social and work participation. Military caregivers (Family Caregivers of wounded or disabled Veterans) reported similar negative effects of becoming a caregiver on their physical and mental health.

Using results from our previous work in mHealth interventions for individuals with SCI, we developed a dual-target intervention for both individuals with SCI and their caregivers.

The overall objective of this research study is to conduct translational research focused on adapting and tailoring the interactive Mobile Health and Rehabilitation (iMHere) 2.0 system to meet the needs of Veterans with SCI and their family caregivers, expanding the psychosocial intervention, and evaluating the feasibility of implementing the iMHere system among Veterans with SCI and their family caregivers.

DETAILED DESCRIPTION:
The overall objective of this project is to conduct translational research focused on adapting and tailoring the iMHere 2.0 system to meet the needs of Veterans with SCI and their FCGs, expanding the psychosocial intervention, and evaluating the feasibility of implementing the iMHere system among Veterans with SCI and their Family Caregivers (FCGs). The specific aims of this project are:

Aim 1: To adapt and tailor the iMHere 2.0 system through a codesign process specifically tailored to meet the needs of Veterans with SCI and their FCGs.

The iMHere 2.0 system was designed for the general population of individuals with SCI, spina bifida, and cerebral palsy age 12 through adulthood. "Codesign" refers to a participatory approach to designing solutions in which participants are treated as equal collaborators in the design process. Codesign means designing with, not for, the participants (Veterans with SCI and their FCGs).

Aim 2: To refine and co-develop the psychosocial dual-target intervention model within iMHere 2.0 to cater specifically to Veterans with SCI and their FCGs.

We have conducted preliminary work on psychosocial interventions both for caregivers and care recipients. In this aim, we plan to expand the existing interventions by combining the materials that have been developed in the previous projects with co-design process of Aim 1 to achieve a user-centered, dual-target intervention that meets the needs of Veterans with SCI and their FCGs.

Aim 3: To conduct a study to evaluate usability and feasibility of implementing the iMHere 2.0 system among Veterans with SCI and their caregivers.

We plan to implement the adapted and expanded iMHere 2.0 system (the result of Aims 1 and 2) among Veterans with SCI and their FCGs in a consumer model of delivery. This includes a variety of care models where iMHere can be implemented: medical, community based, and consumer. In a consumer model, Veterans with SCI and their FCGs will use the iMHere system as a consumer tool outside the medical system.

ELIGIBILITY:
Inclusion Criteria:

* Veterans with SCI or Family caregivers of Veterans with SCI
* Have access to the Internet and a computer to participate in a Zoom call
* Able to speak and understand English to provide informed consent.

Exclusion Criteria:

* Serious mental illness requiring psychiatric hospitalization

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Participants can reside anywhere in the US because the study is conducted remotely via Zoom.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2025-12-01 (Actual); Primary Completion 2029-11 (Estimated); Study Completion 2029-11 (Estimated)

PRIMARY OUTCOMES:
Ratio of actionable feedback to system integration | From enrollment to end of study completion approximately 6 months
  The study will collect actionable feedback and the needs of veterans with SCI and their family caregivers and implement them into the iMHere Mobile Health App system. We will measure the ratio between actionable feedback and needs of veterans with SCI and their family caregivers to the system integration.

SECONDARY OUTCOMES:
Participant Satisfaction | At the end of study participation approximately 6 months after enrollment
  This is a qualitative data, no quantifiable metric(s) will be used. We will gather participants' satisfaction of the result of the codesign process to evaluate how well the implementation of the actionable feedback reflects the perspective and needs of veterans with SCI and their caregivers. This outcome will be collected using interviews that includes questions about usability, acceptability, and utilization of the system. The interview will also identify barriers and facilitators of the iMHere adoption by Veterans with SCI and their family caregivers.

CONTACTS AND LOCATIONS:
Overall Officials: Bambang Parmanto, Ph.D, Study Director — University of Pittsburgh; Yong Choi, PhD, MPH, Principal Investigator — University of Pittsburgh
Locations (1):
- University of Pittsburgh, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Undecided
Data may be shared with other researchers in an aggregate and de-identified manner